CLINICAL TRIAL: NCT04841590
Title: Effects of Osteopathic Manual Therapy on Infant Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, David Nuñez Fernandez, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 380263
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Colic, Infantile
MeSH Terms: conditions — Colic | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental clinical trial will be conducted where the evaluator and parents will be blinded to the allocation group for each subject
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The evaluator will be blinded. Parents will be blinded to the allocation group to which each subject belongs until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group (EG) will receive treatment through the use of manual physiotherapy techniques such as mobilization techniques in the spinal column, cranial techniques and visceral mobilization applied by gentle pressure, according to the therapist's diagnostic criteria after performing palpatory and mobility tests.
  Interventions: Other: Intervention of the experimental group (EG)
- Control Group (Sham Comparator): The control group (CG) will not receive any treatment
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Other: Intervention of the experimental group (EG) — Treatment through the use of manual physiotherapy techniques such as mobilization techniques in the spinal column, cranial techniques and visceral mobilization applied by gentle pressure, according to the therapist's diagnostic criteria after performing palpatory and mobility tests.
  Arms: Experimental Group
Other: Control Group (CG) — Subjects in the control group (CG) will not receive any treatment
  Arms: Control Group

SUMMARY:
Infant colic (CL) is a common disorder that affects approximately 8-33% of newborns during the first months of life. Typically defined as "crying that lasts at least 3 hours a day, and occurs at least 3 days a week over a 3-week period." Osteopathic manual therapy is presented as an effective and safe alternative to CL treatment.

The main objective of the study is to quantify possible changes in daily crying hours and hours of sleep, the severity of CL, the frequency of episodes, changes in stool and possible adverse effects.

The study hypothesis argues that the application of osteopathic manual therapy in babies with CL produces an improvement in the hours of daily crying, the frequency of episodes, the severity of colic and the hours of sleep. A controlled RCT will be performed where the evaluator and the parents will be blinded with respect to the allocation group for each subject. Subjects who meet the inclusion and exclusion criteria will be randomly assigned to the experimental group (EG) and control group (CG) using a table of random numbers by a person from outside the research. The EG diagnosis treatment using techniques of osteopathic manual therapy, vertebral mobilization, cranial techniques and visceral mobilization, according to the diagnostic criteria of the therapist. The CG has no treatment.

A total of 3 procedures were performed, one per week, problems with the chronology in all groups (days 0, 7 and 14 if required).

The therapist in charge of performing the operations will be a Physiotherapist and Osteopath with more than 10 years of experience.

The evaluations will be carried out by a healthcare professional with more than 10 years of experience. The evaluator will be blinded. Parents blinded with respect to the allocation group of each subject until the end of the study.

To analyze the main variable of the study (total hours of excessive crying per day), use the crying diary completed by the parents. The Infantile Colic Severity Questionnaire (ICSQ) will be applied to evaluate the secondary variables (sleep, feces, frequency of episodes and severity of colic).

ELIGIBILITY:
Inclusion Criteria:

* Inconsolable crying for more than 3 hours a day, at least 3 days a week for at least 3 weeks.
* Age 2 - 12 weeks.
* Gestation equal to or greater than 38 weeks.
* Birth weight equal to or greater than 2,500 grams.
* Weight gain of at least 150 grams. per week.
* Appropriate pediatric general physical examination (height, weight, head circumference and psychomotor development).
* Sign the informed consent.

Exclusion Criteria:

* Signs and / or symptoms of other pathologies.
* Signs of lactose intolerance.
* Having had benefits with the withdrawal of milk from maternal feeding or the use of milk with hydrolyzed casein.
* Having received the subjects and / or siblings, previous treatment with Osteopathy and / or Chiropractic.
* Contraindication to the treatment and / or some of its techniques; presence of congenital malformations.

Ages: 2 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Total hours of crying per day | At the beginning of the study (pre-intervention)
  A crying diary completed by the parents will be used to compute the total hours per day that the subject presents crying.
Total hours of crying per day | 1 week after the first intervention
  A crying diary completed by the parents will be used to compute the total hours per day that the subject presents crying.
Total hours of crying per day | 2 weeks after the first intervention
  A crying diary completed by the parents will be used to compute the total hours per day that the subject presents crying.
Total hours of crying per day | 3 weeks after the first intervention
  A crying diary completed by the parents will be used to compute the total hours per day that the subject presents crying.
Total hours of crying per day | Finally at 4 weeks from the first intervention
  A crying diary completed by the parents will be used to compute the total hours per day that the subject presents crying.
Frequency of episodes | At the beginning of the study (pre-intervention), 1 week after the first intervention, 2 weeks, 3 weeks and finally at 4 weeks from the beginning of the study
  The total number of crying episodes per day will be assessed using the Crying Diary completed by the parents.
Frequency of episodes | 1 week after the first intervention
  The total number of crying episodes per day will be assessed using the Crying Diary completed by the parents.
Frequency of episodes | 2 weeks after the first intervention
  The total number of crying episodes per day will be assessed using the Crying Diary completed by the parents.
Frequency of episodes | 3 weeks after the first intervention
  The total number of crying episodes per day will be assessed using the Crying Diary completed by the parents.
Frequency of episodes | Finally at 4 weeks from the first intervention
  The total number of crying episodes per day will be assessed using the Crying Diary completed by the parents.

SECONDARY OUTCOMES:
Colic Severity | At the beginning of the study (pre-intervention), 1 week after the first intervention, 2 weeks, 3 weeks and finally at 4 weeks from the beginning of the study
  Severity will be assessed using the Infantile Colic Severity Questionnaire (ICSQ), a reliable and validated questionnaire for the diagnosis and evaluation of infant colic.
  The numerical values assigned to the responses suppose a score for each item that varies between 1-4 points, where 1 indicates "less seriousness" and 4 "more serious". The total score of the questionnaire is obtained by adding the value achieved in each item, which can range from 24 to 100 points.
Hours of sleep | At the beginning of the study (pre-intervention), 1 week after the first intervention, 2 weeks, 3 weeks and finally at 4 weeks from the beginning of the study
  The total number of hours of sleep will be measured using the Infantile Colic Severity Questionnaire (ICSQ)
Stool | At the beginning of the study (pre-intervention), 1 week after the first intervention, 2 weeks, 3 weeks and finally at 4 weeks from the beginning of the study
  Possible changes regarding this variable will be evaluated using the Infantile Colic Severity Questionnaire (ICSQ), a reliable and validated questionnaire for the diagnosis and evaluation of infant colic.
  The numerical values assigned to the responses suppose a score for each item that varies between 1-4 points, where 1 indicates "less seriousness" and 4 "more serious". The total score of the questionnaire is obtained by adding the value achieved in each item, which can range from 24 to 100 points.
Use of drugs | At the beginning of the study (pre-intervention), 1 week after the first intervention, 2 weeks, 3 weeks and finally at 4 weeks from the beginning of the study
  It will be evaluated if the subjects take drugs at the beginning of the study, as well as the possible changes regarding this variable during the course of the study, using the Crying Diary completed by the parents.

CONTACTS AND LOCATIONS:
Overall Officials: David Nuñez Fernandez, PT, MsC, Principal Investigator — University of Seville
Locations (3):
- Spain (3):
  - Clinica de Fisioterapia y Osteopatía M4, Granada, Granada
  - Hospital del Sureste, Madrid, Madrid
  - Fisioterapia y Osteopatía David Nuñez, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No